CLINICAL TRIAL: NCT06050304
Title: Descriptive Study of Observed Behavioural Awareness and Patients Expectations of Treatment
Brief Title: CRACK-TARGET 1: Descriptive Study of Observed Behavioral Sensitization and Expectations
Acronym: CRACK-TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-A02072-41
Record Dates: First submitted 2023-05-15; First posted 2023-09-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-06

CONDITIONS: Cocaine Use Disorder
Keywords: Crack-cocaine; Behavioral Sensitization
MeSH Terms: interventions — Behavior Observation Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Crack-cocaine Use Disorder users (Experimental): Observation of behaviour in ecological conditions in patients with crack-cocaine dependence
  Interventions: Behavioral: Observation of behavior and search of biomarkers with 3 blood tests.3 weeks wearing an actimeter; Biological: 3 blood tests

INTERVENTIONS:
Behavioral: Observation of behavior and search of biomarkers with 3 blood tests.3 weeks wearing an actimeter — In the form of a small watch, which collects the level of motor activity throughout the day and night. Patients will be asked to indicate each moment of crack-cocaine use by pressing the button in the center of the watch. We want to know if certain uses lead to more behavioral problems (especially after periods of cessation).
Biological: 3 blood tests — We will try to identify biomarkers of BS: blood proteins, genetic markers passed on by your parents, or the expression of proteins in particular situations

SUMMARY:
This research focuses on behavioral sensitization (BS) a specific behavioural disturbance in crack-cocaine addiction. The primary objective is to observe whether BS can be demonstrated in an ecological setting in crack dependent users by continuous actimetry for 3 weeks.

It is planned to include 20 persons with a current crack-cocaine addiction with a preferential use of rapid administration route (intravenous or smoke), in a care institution: Fernand Widal Hospital.

In the proposed research, the investigators will assess the movements of crack-cocaine dependent users in relation to consumption. They will have to wear continuously for 3 weeks an actimeter. They will also have 3 blood tests trying to identify biomarkers of BS.

DETAILED DESCRIPTION:
Paris region and the French west indies face a specific epidemic of crack-cocaine use, mostly by socially deprived subjects, highly visible in open drug scenes, with little access to the care system. Patients who suffer from crack-cocaine dependence experiment a high rate of medical and a high mortality rate, because this type of cocaine is a short-acting form, used through rapid route of administration (usually smoked or injected).

Nevertheless, despite important uncovered medical needs, they are not often included in clinical trials and there is to date no pharmacological treatment for this severe condition. The investigators identified behavioral disturbances as a key problem in crack-cocaine dependence, as it is the second cause for emergency visits for those patients and a reason to be excluded from addiction care facilities.

Based on preliminary results already gathered by our group, the investigators suggest that behavioral sensitization (BS), an increase of motor response to cocaine after repetitive intermittent use, could be assessed in Humans.

Our goal is therefore to include 20 persons (10 males - 10 females) with a current cocaine use disorder,specifically crack users, with preferential use of rapid administration route (intravenous or smoke), in a care institution: the Fernand Widal Hospital (Assistance Publique - Hôpitaux de Paris). The investigators will assess the movements of crack-cocaine dependent users in relation to consumption. They will have to wear continuously for 3 weeks an actimeter, in the form of a small watch, which collects the level of motor activity throughout the day and night. They will be asked to indicate each moment of crack-cocaine use by pressing the button in the center of the watch. The investigators want to know if certain uses lead to more behavioral problems (especially after periods of cessation).

They will also have 3 blood tests: the investigators want to know if blood proteins, genetic markers passed on by paricipants parents or the expression of proteins in particular situations, could predict this increase in motor effects for small doses of crack-cocaine.

The investigators also want to better understand the needs of crack-cocaine dependent patients towards treatments and their expectations for recovery, by conducting a qualitative study where patients will participate in the definition of treatment aims to increase the efficiency of care

With the project CRACK-TARGET 1 : DETA, the investigators aim at demonstrating the existence of BS in patients with crack dependent subjects. Furthermore, the investigators aim at developing specific, repeatable, easy to access measure of BS using questionnaires and objective actigraphy biomarkers to be used as surrogate endpoints in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Have a current crack-cocaine use disorder defined as Severe Intensity Use Disorder (6 or more DSM5 criteria), AND preferential use of rapid administration route (intravenous or smoked)
* Self-identified male or female (n=10 males, n=10 females)
* Negative pregnancy test for females and use of effective contraception
* Be affiliated with a social security plan (or PUMA or CSS or AME)
* Sign an informed consent and commit to a 3-week follow-up in the study
* Have a weight greater than 40 kg

Exclusion Criteria:

* • Patient with a psychiatric disorder or symptoms that are not currently stabilized

  * Patient who is a minor or under protective supervision (curatorship or guardianship)
  * Patient in care at the request of a judicial authority (therapeutic injunction, classification with orientation)
  * Pregnant or breastfeeding women
  * Patients who do not speak French or English sufficiently
  * Patients weighing less than 40 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Crack-Cocaine Use Disorders patients, men and women
Enrollment: 20 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-03-04 (Estimated); Study Completion 2026-03-04 (Estimated)

PRIMARY OUTCOMES:
Reduction in sleep duration(hours/minutes) on crack-cocaine use days following a break of at least 2 days compared to crack-cocaine use days without any break (means over the 3 weeks period) | 3 Weeks
  Reduction in sleep duration(hours/minutes) on crack-cocaine use days following a break of at least 2 days compared to crack-cocaine use days without any break (means over the 3 weeks period)

SECONDARY OUTCOMES:
Earlier onset of M10(the time of day when the 10 hours of peak motor activity begins, a reflection of the "motor wake-up time). | 3 Weeks
  The time of day when the 10 hours of peak motor activity begins, a reflection of the "motor wake-up time") (hours/minutes) during crack-cocaine use days following a 2 days break compared to crack-cocaine use days without any break (comparison of mean M10 time)
Shorter relative amplitude of motor activity (the relative difference between M10) | 3 Weeks
  Average activity level during the most active 10-hour period) and L5 (average activity level during the least active 5-hour period) (hours/minutes) during crack-cocaine use days following a 2 days break compared to crack-cocaine use days without any break (comparison of mean relative amplitudes over 3 weeks
Self-defined patients' expectations toward treatment measured in qualitative interviews | 3 Weeks
  Expectations toward treatment measured in qualitative interviews
Higher scores assessed with questionnaires that approximate BS | 3 weeks
  Higher scores assessed with questionnaires that approximate BS
WURS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS | 3 weeks
  WURS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS
ASRS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS | 3 weeks
  ASRS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS
SAPS-CIP in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS | 3 weeks
  SAPS-CIP in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS
YMRS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS | 3 weeks
  YMRS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS
UPPS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS | 3 weeks
  UPPS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS
PDI in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS | 3 weeks
  PDI in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS
PANSS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS | 3 weeks
  PANSS in patients presenting with at least 1 of the 3 previously defition of BS on actimetric measures compared to patients without BS

OTHER OUTCOMES:
A/G % in rs7568970 polymorphism of the LRP1B gene in patients with observed versus without observed BS | 3 weeks
  Fold change of the methylation status of the LRP1B gene in patients with observed versus without observed BS

CONTACTS AND LOCATIONS:
Overall Officials: Florence VORSPAN, Principal Investigator — Hôpital Fernand Widal
Locations (2):
- France (2):
  - Centre 001_Hôpital Fernand Widal, Paris
  - Hôpital Fernand Widal, Paris

IPD SHARING:
Plan to Share IPD: Yes
IPD can be available upon reasonable request made to the promotor (DRCI APHP)